CLINICAL TRIAL: NCT02981329
Title: Use of Metformin as a Fetal Hemoglobin Inducer in Patients With Hemoglobinopathies
Brief Title: Fetal Hemoglobin Induction Treatment Metformin
Acronym: FITMet
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Titilope Fasipe, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-38457 Metformin
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Sickle Cell Anemia; Sickle Cell Disease; Hemoglobin Disorder
Keywords: Metformin; Sickle Cell Anemia; Sickle Cell Disease; Hemoglobinopathies; Hemoglobin Disorder; Blood Disease; Hemoglobin Disease
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobinopathies; Hematologic Diseases | interventions — Metformin; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: Hydroxyurea + Metformin (Experimental): Subjects who are currently taking Hydroxyurea as part of standard of care and have sickle cell anemia.
  Interventions: Drug: Metformin; Behavioral: Questionnaires
- Group B: Metformin (Group B has closed to enrollment) (Experimental): Subjects who are not taking Hydroxyurea as part of standard of care and have sickle cell anemia.
  Interventions: Drug: Metformin; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Metformin — Metfomin will be taken daily. The metformin dose will be increased during two time points per subject if protocol dose escalation criteria is met.
  Other Names: Glucophage; Riomet,
Behavioral: Questionnaires — Questionnaires will be completed to assess the impact quality of life

SUMMARY:
The purpose of this study is to determine whether metformin is effective in the treatment for sickle cell anemia (SCA).

DETAILED DESCRIPTION:
This is a dose escalation, pilot study for subjects with sickle cell anemia (SCA) disease to determine if metformin has a beneficial effect on the treatment and quality of life of SCA patients.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of sickle cell anemia
2. Age greater than or equal to 10 and less than or equal to 60 years of age.
3. If on hydroxyurea, fetal hemoglobin less than 20% at a stable dose (mg/kg) determined by the primary hematology provider over at least four months.
4. Creatinine less than or equal to 1.4 mg/dL and estimated glomerular filtration rate greater than 45 ml/min/1.73 m2
5. Liver function tests (specifically ALT and conjugated bilirubin) less than or equal to 4 times upper limits of normal.

Exclusion Criteria:

1. Failure to meet inclusion criteria
2. Simple or chronic red blood cell transfusion therapy in the last 3 months OR a HbA level greater than 5% in SCA patients
3. Refusal to use medically effective birth control if female and sexually active.
4. If on hydroxyurea, not at stable dose of hydroxyurea for a minimum of 4 months (temporary exclusion).
5. Creatinine greater than 1.4mg/dL
6. Liver function tests (ALT and conjugated bilirubin) greater than 4 times upper limits of normal.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Change in Fetal Hemoglobin (HbF) Percentage (SCA) or Change in Total Hemoglobin (Hb) | 1 Year
  Change in HbF percentage (%) or total Hb will be assessed by comparing baseline values to on treatment values per subject and will be summarized.

SECONDARY OUTCOMES:
Change in Laboratory Values | 1 Year
  Evaluation and percentage of change in numeric values of total blood count, liver function, HbF levels, whole blood viscosity, and percent dense red blood cells will be evaluated per subject over the duration of the study and summarized.
Impact on Quality of Life | 1 Year
  Evaluation of subject's change in quality of life will be assessed per subject per study questionnaire(s) over the duration of the study and summarized.
Variability of Hemoglobin Response | 1 Year
  Evaluation of hematological variability of fetal hemoglobin induction will be assessed per subject per genetic analysis and summarized.
Evaluation of RNA Sequencing | 1 Year
  Evaluate expression changes in paired samples collected before and on metformin through RNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Titilope Fasipe, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The leftover blood samples for genetic analysis will be banked indefinitely for future ancillary studies. Investigator who desires access to these samples must present their research idea prior to receiving access to the samples. The samples will be shared with researchers affiliated with Texas Children's Hospital, Baylor College of Medicine and/or other hematology collaborators for future studies associated with hematologic diseases and drugs used to treat such diseases. The recipient investigators are required to provide proof of IRB approval or exemption as per local IRB guidelines before the sample can be released for research purposes. After receipt of IRB approval, coded samples will be distributed to the recipient investigator.